



# **Research Proposal Form**

| This section is for Official Use Only | | |
|---|---|---|
| Reference Code: | Date of application (dd/mm/yyyy): | |
| This section is for the applicant to fill. Lucy Times New Pomens Font, size 11 and adjust 1 | lina snaoina ta | 1.5 all through the application form |
| <ul> <li>Use Times New Romans Font, size 11 and adjust line spacing to 1.5 all through the application form</li> <li>Do not CAPITALIZE all words</li> </ul> | | |
| Part 1: General | | |
| Tart 1. General | _ | |
| Master Degree b. MD | c. Iı | ndependent Research/Project |
| <b>1.1 Applicant Name</b> (responsible for all correspondences | and accuracy of | f data): Department: |
| Maikel Merit Gerges Morkos | | General surgery |
| e-mail address: Michael.16266363@med.aun.edu.eg Mobile Phone: 01271267725 | | |
| ة :مایکل مریت جرجس مرق <i>س</i> | الاسم باللغة العربيا | Home Phone: 01091018115 |
| 1.2 English Title of research project: | | |
| Role of Platelet Rich Plasma in Bone regeneration after e | nucleation of od | dontogenic jaw cysts |
| <b>1.3 Arabic Title</b> (use the WHO Unified Medical Dictional | ary)• www.emro | who int/unified_madical_dictionary.html |
| · · | • / | دور البلازما الغنية بالصفائح الدموية في تجديد العظا |
| | ., - 0 | , · <b>G</b> .5 C · · · · 5 · 55 |
| 1.4 Do you need funding from Assiut Medical Scho | ol Grants Offic | ce? |
| Yes No | | |
| Mention other sponsoring agent(s) if any: | | |
| 1 | | |
| Assiut Medical School Research Proposal Form | | |





#### Part 2: Research Details

**2.1 Background** (Research Question, Available Data from the literature, Current strategy for dealing with the problem, Rationale of the research that paves the way to the aim(s) of the work). (200-250 words max.)

Jaw cysts are common lesions in the oral and maxillofacial region. Enucleation of cyst wall & curettage has evolved as the treatment of choice. In order to reduce infections and to accelerate bone regeneration, by using of Platelet rich plasma.

Platelets are involved in regeneration at sites of pathology, apart from their role in clotting. A preparation composed mainly of platelets (platelet-rich plasma gel)

applied to sites of bony pathology, after surgical treatment of lesions, may hasten bone regeneration.

An interesting idea developed that the addition of a concentrate of platelets, to wounded tissues or surgical sites, may enhance the body's natural wound healing mechanisms [1]. Platelet-rich plasma (PRP) is the accepted term to describe the preparation made out of autologous platelets suspended in autologous plasma, in concentration greater than normally found in peripheral blood

Because it is autologous, PRP avoids the risk of transmissible diseases such as HIV, Hepatitis B, C or D and other blood-borne pathogens [2]. A clot accelerator such as bovine thrombin is added to gel the PRP or PRP is added to other materials such as collagen, gelfoam, etc.

#### 2.2 Aim(s) of the Research (50 words max):

in the present study, the effect of PRP on bone regeneration when applied to the site of removal of cyst of the jaws is evaluated. PRP was delivered to the site combined with gelfoam. Thrombin clot accelerator was not used.

#### 2.3 Research Domain (Faculty Research Plan).

- 1. **Trauma**; epidemiology, prevention, management, and rehabilitation
- 2. Communicable diseases; prevention, screening for early detection, and management
- 3. **Infection** control and health-care-associated infections and Safety of medical service providers
- 4. **Population** problem, maternal and perinatal morbidity and mortality
- 5. **Non-communicable diseases**; prevention, screening for early detection, and management
- 6. **Evidence based management** of common medical and surgical problems
- 7. Organ Transplantation
- 8. **Geriatric Health**; promotive, preventive, curative and rehabilitative services
- 9. Stem cells and/or tissue culture application in managing various diseases in clinical trials
- 10. **Experimental Research**; basic and animal model research that may lead to possible enhancement in health services
- 11. Others, clarify,-----

#### 2.4. Research Methods and techniques:

# The state of the s

## Faculty of Medicine Institutional Review Board (IRB)



- 2.4.1- Type of the study: interventional, prospective clinical trials
- 2.4. 2- Study Setting: general surgery department , Assiut university , in the period from 10/2024 to 10/2026

#### 2.4. 3- Study subjects:

#### a. Inclusion criteria:

- 1. All patients admitted to AUH with mandibular or maxillary Odontogenic cysts
- 2. Size of the cyst more than 2 cm
- 3. The lesion could be visualized radiographically
- 4. Patients within the age range of 20 to 50 years

#### b. Exclusion criteria:

- 1-Neoblatic lesions
- 2- Patients who were alcoholics & smokers
- 3-Patients with systemic diseases
- 4-History of bleeding tendencies, blood dyscrasia
- 5-Low platelet count
- 6- Patients unable or unwilling to return for follow-up
- **c. Sample Size Calculation:** The sample size was calculated using G\*power software 3.1.9.4., the minimum required sample size is 42 patients (21 in each group)

based on the

following assumptions:

The main outcome variable is the role of Platelet Rich Plasma in Bone regeneration after enucleation of odontogenic jaw cysts. Based on previous study (Evaluating the Efficacy of Platelet-Rich Plasma (PRP) in Accelerating Healing and Reducing Complications in Oral Surgery) we expect to find large effect size = 1 164

The main statistical test is t-test to detect the difference between the two groups.

Two tailed

Alpha = 0.05

Power = 0.95

Effect size = 1.164

Allocation ratio= 1

The Parameters:





Mean  $\pm$  SD of The alveolar bone density in PRP

patients at 6 months postoperative: 141.13±10.81

Mean  $\pm$  SD of control group at 6 months postoperative : 127.91 $\pm$ 11.87

#### 2.4.4 – Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, ...):

#### • Patient history

history of tooth extraction pain in jaw

#### Examination

jaw or maxillary swelling

#### Laboratory investigation

Complete blood picture

Coagulation profile

Kidney function

Liver function

#### Imaging

panorama xray

CT teeth

#### Instruments & method

#### Preparation of PRP

Preoperatively, platelet-rich plasma was prepared in the Haematology Laboratory from 20 ml of the patient's blood using an R8-C Laboratory Centrifuge (Remi Motors Ltd., Mumbai) using an aseptic technique.

#### Armamentarium

Anticoagulant citrate phosphate dextrose, sterile 10 ml test tubes (2 nos.), sterile pipette, Vacutainer tubes 5 ml (2 nos.), 10 ml syringe and 21 gauge needle were used.

#### **Procedure**

Twenty millilitres of venous blood is collected from antecubital region with a 20- ml syringe and transferred to two test tubes containing 1.4 ml anticoagulant (citrate phosphate dextrose solution) each. (A ratio of 1.4 ml of anticoagulant to 10 ml of blood) It is then centrifuged for 10 min at 1,300 rpm. The result is a separation of whole blood into a lower red blood cell region and an upper straw colored plasma region

#### Surgical procedure





The enucleation of cyst or tumour and any further treatment to eliminate pathology was performed nder local anesthesia, or in case of large lesions, treatment was performed under general anesthesia. Affected teeth were either removed or treated endodontically.

In the study group, for Mlling the bony defect PRP gel was used. At the time of application, 1 ml of  $10\,\%$  calcium gluconate was added to the PRP and mixed well. A small cube of Gelfoam was added to the test tube to soak load PRP (Fig. 4). The test tube

was left standing for 5 min. A gel formed that was placed inside the defect . Primary wound closure was performed.

**Postoperative follow-up:** after one month, three months & six months

#### 2.4.5 – Research outcome measures:

a. Primary (main):

1 infection

2.bone healing

b. Secondary (subsidiary):

1 operation time

2 hospitalization time

3 Recurrence

#### 2.5-Data management and analysis (Details needed):

**Data collection**: data will be collected in patient sheet.

**Computer software**: Microsoft Office, SPSS statistical program

**Statistical tests:** Data will be managed by Microsoft Excel, Statistical analysis of the data will be Performed using SPSS\_22 software package, Data will be presented in the form of frequency and percent, Studied groups will be evaluated by analysis of variances.

# 2.6-References (max. 15) and written in Vancouver style:

- 1. Doiphode AM, Hegde P, Mahindra U, Santhosh Kumar SM, Tenglikar PD, Tripathi V. Evaluation of the efficacy of platelet-rich plasma and platelet-rich fibrin in alveolar defects after removal of impacted bilateral mandibular third molars. J Int Soc Prevent Communit Dent 2016;6:S47-52.
- 2. Hanif M, Sheikh MA. Efficacy of platelet rich plasma (PRP) on mouth opening and pain after surgical extraction of mandibular third molars. J Oral Med Oral Surg 2021;27:9.
- 3. Tiwari A, Gupta N, Singla D, Swain JR, Gupta R, Mehta D, et al. Artificial intelligence's use in the diagnosis of mouth ulcers: A systematic review. Cureus 2023;15:e45187. doi: 10.7759/cureus.45187.
- 4. Intini G. The use of plateletrich plasma in bone reconstruction therapy. Biomaterials 2009;30:4956-66.





- 5. Tiwari A. A traumatic ulcer caused by accidental lip biting following topical anesthesia: A case report. Cureus 2023;15:ee38316. doi: 10.7759/cureus.38316.
- 6. Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, et al. Plateletrich fibrin (PRF): A secondgeneration platelet concentrate. Part I: Technological concepts and evolution. Oral Surg Oral Med Oral Pathol Oral Radiol Endod 2006;101:e37-44.
- 7. Tiwari A, Kumar A, Jain S, Dhull KS, Sajjanar A, Puthenkandathil R, et al. Implications of ChatGPT in public health dentistry: A systematic review. Cureus 2023;15:e40367. doi: 10.7759/cureus.40367.
- 8. Rathore A, Tiwari A, Nazim M, Gupta AK, Gande M, Krishnakumar J. Detection of human papillomavirus and its association with potentially malignant disorders and oral squamous cell carcinoma: A retrospective study. J Pharm Bioallied Sci 2022;14(Suppl 1):S820-4.
- 9. Kulkarni MR, Thomas BS, Varghese JM, Bhat GS. Plateletrich fibrin as an adjunct to palatal wound healing after harvesting a free gingival graft: A case series. J Indian Soc Periodontol 2014;18:399-402.

# Part 3: Ethical Considerations (Written in detail taking into consideration the items below):

#### 3.1. Risk – benefit assessment:

As the study is observational, there are no additional risks to the patients other than the recognized risks of their standard care.

3.2. Confidentiality (dealing with data and data dissemination should be confidential).

The confidentiality of all participants admitted to this study will be protected to the fullest extent possible. The study participants will not be identified by name in any report or publication resulting from data collected in this study.

3.3. Statement describing the research procedure to be given to the participants.

Ethical aspects whether substantial or procedural will be implicated in this study. Before participants are admitted in this study, the purpose and nature of the study as well as the risks will be explained to their parents. The participants and/or their parents must agree that he/she understands the investigational nature of the study, its inherent risks and benefits, his/her rights to terminate participation in this study without affecting his/her rights in having proper health care in the study site, whom to contact with questions regarding the study and that he/she is freely given an informed consent to participate in this study

3.4. Informed consent.

Informed written or oral consent of the patients will be acquired before participation in the study.

- 3.5. Other ethical concerns:
  - The research should be conducted only by scientifically qualified and trained personnel.
  - The research should be based on relevant pre-clinical investigations in animals.
  - The detailed consent form must be inserted here in the proposal.

إقرار بالموافقة على المشاركة في البحث





| | | اقر انا |
|---|---|---|
| بانني اطلعت على بيان مفصل عن البحث المقدم من الطبيب طم /مايكل مريت جرجس مرقس | | |
| وانه قد تم اطلاعي على الهدف من هذه الدراسة واستراتيجية الدراسة كاملة كما وردت في استراتيجية البحث مع ذكر احتمالات المتاعب | | |
| التي قد يرد حدوثها من الدراسة وانه سوف لا يترتب على عدم موافقتي على الاشتراك في البحث حجب اي خدمة طبيه عني | | |
| ، لى الفرصة السؤال عما اريد وتم اجابة اسئلتي جميعها وبما ارضاني | المعلومات السابقة او قرئت عليا وكانت | لقد قرات |
| دراسة و افهم انه من حقى التوقف عن المشاركة فيها في اى وقت لاحق دون أن يؤثر ذلك | كامل اختياري على المشاركة في هذه الد | واوافق بك |
| على الخدمة الكلية المقدمه لي | | |
| | ريض المشارك في البحث | توقيع المر |
| | | العنوان |
| | | التاريخ |
| Part 4: Funding (Mandatory for those requesting funding from | om Grant Office) | |
| | · | |
| 4.1. Total funds requested: LE | | |
| 4.2. Author responsible for managing the budget/grant (Cannot be a | 4.2. Author responsible for managing the budget/grant (Cannot be a resident): | |
| Name | | |
| Name Department | · | |
| Name | · | |
| Name Department e-mail Mol | pile | |
| Name Department e-mail 4.3. Budget Details | · | |
| Name Department e-mail Mol 4.3. Budget Details Research equipment and accessories | pile | |
| Name Department e-mail 4.3. Budget Details Research equipment and accessories Chemicals/Medications | pile | |
| Name Department e-mail Mol 4.3. Budget Details Research equipment and accessories | pile | |
| Name Department e-mail 4.3. Budget Details Research equipment and accessories Chemicals/Medications | pile | |
| Name Department e-mail 4.3. Budget Details Research equipment and accessories Chemicals/Medications Data entry | pile | |
| Name Department e-mail 4.3. Budget Details Research equipment and accessories Chemicals/Medications Data entry | pile | |
| Name Department e-mail 4.3. Budget Details Research equipment and accessories Chemicals/Medications Data entry Statistical analysis 4.4. All researchers' International publications in the last 3 years. | Dile | Impact |
| Name Department e-mail 4.3. Budget Details Research equipment and accessories Chemicals/Medications Data entry Statistical analysis 4.4. All researchers' International publications in the last 3 years. Title | pile | Impact<br>Factor |
| Name Department e-mail 4.3. Budget Details Research equipment and accessories Chemicals/Medications Data entry Statistical analysis 4.4. All researchers' International publications in the last 3 years. Title Title | Dile | - |
| Name Department e-mail 4.3. Budget Details Research equipment and accessories Chemicals/Medications Data entry Statistical analysis 4.4. All researchers' International publications in the last 3 years. Title | Dile | - |





(Add others if required)

# 4.5. Details of Previously Obtained Grants (institutional or others):

| | Title | Name of<br>Applicant for<br>grant | Date<br>obtained | Finished<br>Yes/No | Published<br>Yes/No |
|---|---|---|---|---|---|
| 1 | | | | | |
| 2 | | | | | |
| 3 | | | | | |
| 4 | | | | | |

(Add others if required)





# 4.6. Research reporting timetable (Mandatory if applying for a fund):

| Activity (Other activities may be added) | Time required (Months) | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20 | 22 | 24 |
| Preparation and development of Material | | | | | | | | | | | |
| Training of personnel involved in the research (if needed) | | | | | | | | | | | |
| Research work (Clinical, lab work or field work) | | | | | | | | | | | |
| Data entry and analysis | | | | | | | | | | | |
| Research writing | | | | | | | | | | | |
| Publication | | | | | | | | | | | |

<sup>\*</sup> Numbers indicates the time in months needed to complete each part of the project.

يتعهد الباحثون بنشر نتائج البحث الممول من وحدة تمويل الأبحاث في إحدى الدوريات العلمية المحكمة والمدرجة على قاعدة Scopus أو Web Of Science في خلال الفترة الزمنية المحددة في البند السابق من قبلهم والا يتم خصم مبلغ التمويل من مرتباتهم بالتساوى فيما بينهم كما يتعهدوا بالإشارة الى مساهمة وحدة تمويل الأبحاث بكلية طب أسيوط عند نشر البحث.

<sup>\*</sup> Please half squares corresponding to time required for each specific action





# **Part 5 – Declaration** (Name in printed letters):

I / we (<u>all investigators</u>) certify that, to the best of our knowledge and after reasonable inquiry, the information contained in this application, and any supporting documents provided with this application, are **correct and complete**, and that this research has not been conducted or published before.

يتعهد الباحثون بنشر نتائج البحث الممول من وحدة تمويل الأبحاث في إحدى الدوريات العلمية المحكمة والمدرجة على قاعدة Scopus أو Web Of Science في النوريات النترة الزمنية المحددة في البند السابق من قبلهم والايتم خصم مبلغ التمويل من مرتباتهم بالتساوى فيما بينهم كما يتعهدوا بالإشارة الى مساهمة وحدة تمويل الأبحاث بكلية طب أسيوط عند نشر البحث.

| A | Authorship Responsibility (Add more authors if required) | | | | | | |
|---|---|---|---|---|---|---|---|
| | Title | Name | Role** | e-mail | Phone | Department | Signature |
| 1 | Prof | Samy Mohamed Osman Masoud | 1.1 | samyosman@aun.edu.eg | 0100151964 | General | |
| | | | 2.2 | | 2 | surgery | |
| | | | 3.4 | | | | |
| 2 | Prof | Diaa El-Din Saber Ahmed | 1.3 | dr.diaasaber@gmail.com | 0100796794 | General | |
| | | | 2.1 | | 6 | surgery | |
| | | | 3.1 | | | | |
| 3 | Prof | Ahmed Abdo Gad Yousuf | 1.2 | ahmeddeek2020@aun.edu | 0109710455 | General | |
| | | | 2.2 | .eg | 0 | surgery | |
| | | | 3.3 | | | | |
| 4 | Resi | Maikel Merit Gerges Morkos | 1.2 | Michael.16266363@med. | 0127126772 | General | |
| | dent | | 2.1 | aun.edu.eg | 5 | surgery | |
| | | | 3.1 | | | | |
| 5 | | | | | | | |

<sup>\*\*</sup>Choose at least 1 from each of the 3 groups below





| Group 1 | Group 2 | Group 3 |
|---|---|---|
| 1.1- Conception and design 1.2- Acquisition of data 1.3- Analysis and interpretation of data | 2.1- Drafting of the submitted protocol 2.2-Critical revision of the submitted protocol for important intellectual content | 3.1- Statistical analysis 3.2- Obtaining funding 3.3- Administrative, technical, or material support 3.4- Supervision 3.5- Other (specify) |

#### After completing the application form, please

- 1. Record the completed and revised application form on a CD and present to the Vice Dean Research Office.
- 2. All authors should sign a printed copy of the completed application form that should be presented as well to the Vice Dean Research Office.
- 3. A copy of the printed and signed research application form should be presented to the Ethical Committee.
- 4. It is the applicant responsibility to make sure that the application form is fully and accurately completed and that all other supporting documents or formalities are completed in due time.